CLINICAL TRIAL: NCT05650619
Title: Recurrence Post-transplant Observational Study in Focal Segmental Glomerulosclerosis (FSGS) and Minimal Change Disease (MCD)
Brief Title: Recurrence Post-transplant Observational Study in Focal Segmental Glomerulosclerosis and Minimal Change Disease
Acronym: RESOLVE
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Eloise Salmon, Assistant Professor of Pediatrics, University of Michigan
Other Study IDs: HUM00221259
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Focal Segmental Glomerulosclerosis; Minimal Change Disease; FSGS; MCD
Keywords: Kidney disease; Kidney transplant; Adult; Children; Recurrence
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Nephrosis, Lipoid; Macular dystrophy, corneal type 1; Kidney Diseases; Recurrence | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Optional: DNA bio-specimens blood or saliva.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Enrolled participants prior to transplant: Participants will be consented.
  Interventions: Other: Biospecimen collection; Other: Data collection
- Enrolled participant after transplant: Participants will be consented.
  Interventions: Other: Biospecimen collection; Other: Data collection
- Retrospective participant data: Waiver of consent for secondary use of existing data.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Biospecimen collection — Specimens that may be collected include urine, blood, saliva, kidney tissue, etc. Biospecimens will be collected to establish the RESOLVE biobank.
  Groups: Enrolled participant after transplant; Enrolled participants prior to transplant
Other: Data collection — Data collection for all groups

SUMMARY:
The morbidity of recurrence of focal segmental glomerulosclerosis (FSGS) and minimal change disease (MCD) after transplant is well-recognized and include contemporary reduction in quality of life, edema, early graft loss and mortality. Efforts to understand its mechanisms and improve its treatment have been limited by small sample sizes in single center studies and misclassification in registry studies. Recent advances in the understanding of the mechanisms of FSGS in the native kidney has reinvigorated the scientific community to develop a collaborative community to advance research into the epidemiology, mechanisms, interventions, and outcomes.

The purpose of RESOLVE is to gather a group of people with FSGS and MCD that have had or will have a kidney transplant to create a bank of information and biospecimens so researchers can more effectively study these diseases.

DETAILED DESCRIPTION:
RESOLVE is a multicenter, observational cohort study to examine the post-transplant course of patients with FSGS and MCD across the lifespan. The study is designed to collect both retrospective and prospective data as well as biospecimens and patient reported information. With multiple enrollment options, the study will allow investigators to define the incidence and prevalence of FSGS recurrence, describe the post-transplant course of patients with FSGS and MCD across the lifespan, and develop a biorepository to support future translational research studies to explore relevant disease mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Retrospective non-consented participant group had a transplant from the year 2000 and onward.
* Diagnosis of FSGS or MCD in the native kidney (prior to transplant).

Exclusion Criteria:

* Pathologic diagnosis other than FSGS or MCD
* FSGS or MCD secondary to a known disorder (e.g. lupus nephritis, Immunoglobulin A (IgA) nephropathy, malignancy)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include up to 10,000 subjects across three cohorts. Based on scoping data approximately 250 cases will be available from University of Michigan and approximately 100-350 from each additional participating site.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time to FSGS Recurrence | 2 years after transplant
Time to Graft Failure | 2 years after transplant

SECONDARY OUTCOMES:
Define the Endophenotypes in each group of recurrent FSGS and MCD | 2 years after transplant
  Classifications for the dataset using non-hierarchical clustering techniques
Proportion of recurrence and time to graft failure | 2 years after transplant
Proportion with acute rejection | 2 years after transplant
Proteinuria change over time | Baseline (at transplant), 2 years
Proportion with delayed graft function | 2 years after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Eloise Salmon, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No